CLINICAL TRIAL: NCT02438735
Title: The Effect Of The Presence Of Endometriomas On Ovarian Reserve
Brief Title: Endometrioma Related Reduced Ovarian Reserve
Acronym: ERROR
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, prof.md, Uludag University
Other Study IDs: 2015-7/12
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Endometriosis
Keywords: ovarian endometriomas; AMH; ovarian reserve
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Anti-mullerian hormone (AMH)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Endometrioma: Reproductive aged women diagnosed with endometrioma. Conservative follow up for six months.
  Interventions: Other: Conservative follow up
- Healthy Controls: Women with regular menstrual cycles and without ovarian pathology will be recruited from physicians, nurses and other staff of the same hospital.
  Controls will be matched for age with the women in the endometrioma group. They will be conservatively followed up for six months.
  Interventions: Other: Conservative follow up
- Historical controls who underwent surgical excision: 20 women who underwent surgical excision of endometrioma in the same clinic had serum AMH levels measured preoperatively and on post operative sixth month. Their values will be compared with that of endometrioma group. These data were priorly published in detail (Uncu et al. 2013).
  Interventions: Procedure: laparoscopic endometrioma excision

INTERVENTIONS:
Procedure: laparoscopic endometrioma excision
  Groups: Historical controls who underwent surgical excision
Other: Conservative follow up
  Groups: Endometrioma; Healthy Controls

SUMMARY:
Prior studies have shown surgical excision of endometriomas are associated with a decline in ovarian reserve as assessed by serum anti-Mullerian Hormone (AMH) levels. However, the natural history of serum AMH levels in the presence of untreated endometriomas are unknown. Purpose of this study is to determine whether the presence of endometriomas cause a faster decline in serum AMH levels than in healthy women over a six months period.

DETAILED DESCRIPTION:
The study is a prospective cohort study. Women diagnosed with endometriomas by transvaginal or transabdominal ultrasound or MRI will be recruited from a tertiary care endometriosis clinic. Age matched healthy controls will be recruited from the staff of the same hospital. A priorly published historical group of women who underwent endometrioma excision will be a second comparator.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age
* Endometrioma without indication for surgery or treatment with combined contraceptive, progestin or other hormonal intervention.

Exclusion Criteria:

* Menstrual cycle irregularity
* Polycystic ovarian syndrome
* Women who were pregnant or contemplating pregnancy in the next six months
* History of ovarian surgery
* Using medication which could affect ovarian function during six months before recruitment
* Indication for surgical excision

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The decision to include a healthy control group was taken five months after starting recruitment of women with endometrioma. Only 12 women with endometriomas had been recruited until then and none of them had six month serum AMH level measured.
  Since healthy controls were reluctant to undergo transvaginal ultrasound examination, antral follicle counts were not measured as another marker of ovarian reserve for healthy controls and some women in the endometrioma group.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Serum Anti- mullerian hormone (AMH) level | at recruitment and six months later

CONTACTS AND LOCATIONS:
Overall Officials: gürkan uncu, Study Director — Uludag University School of Medicine
Locations (1):
- Uludag University Scholl of medicine, Bursa, Turkey/bursa, Turkey (Türkiye)

REFERENCES:
- [Background] Uncu G, Kasapoglu I, Ozerkan K, Seyhan A, Oral Yilmaztepe A, Ata B. Prospective assessment of the impact of endometriomas and their removal on ovarian reserve and determinants of the rate of decline in ovarian reserve. Hum Reprod. 2013 Aug;28(8):2140-5. doi: 10.1093/humrep/det123. Epub 2013 Apr 26. PMID 23624580
- [Derived] Kasapoglu I, Ata B, Uyaniklar O, Seyhan A, Orhan A, Yildiz Oguz S, Uncu G. Endometrioma-related reduction in ovarian reserve (ERROR): a prospective longitudinal study. Fertil Steril. 2018 Jul 1;110(1):122-127. doi: 10.1016/j.fertnstert.2018.03.015. Epub 2018 Jun 20. PMID 29935810